CLINICAL TRIAL: NCT06618729
Title: Acute Effects of Plant-based Meat Alternatives Made From Pea, Wheat or Soy Protein in Comparison to Chicken Meat on Postprandial Metabolism in Healthy Women and Men
Brief Title: Effects of Plant-based Meat Alternatives in Comparison to Chicken Meat on Postprandial Metabolism in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Sarah Egert, Prof. Dr. Sarah Egert, University of Bonn
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AlProPlant-HS2
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Plasma Amino Acid Appearance and Disappearance; Postprandial Metabolic Events
Keywords: Postprandial metabolic events
MeSH Terms: interventions — Pea Proteins; Soybean Proteins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pea protein (Experimental): Participants randomized to receive a meal containing 40 g of protein from pea protein extrudate
  Interventions: Other: Pea protein
- Wheat protein (Experimental): Participants randomized to receive a meal containing 40 g of protein from wheat protein extrudate
  Interventions: Other: Wheat protein
- Soy protein (Experimental): Participants randomized to receive a meal containing 40 g of protein from soy protein extrudate
  Interventions: Other: Soy protein
- Chicken (Active Comparator): Participants randomized to receive a meal containing 40 g of protein from chicken meat
  Interventions: Other: Chicken

INTERVENTIONS:
Other: Pea protein — Ingestion of a meal containing 40 g of protein from pea protein extrudate
  Arms: Pea protein
Other: Wheat protein — Ingestion of a meal containing 40 g of protein from wheat protein extrudate
  Arms: Wheat protein
Other: Soy protein — Ingestion of a meal containing 40 g of protein from soy protein extrudate
  Arms: Soy protein
Other: Chicken — Ingestion of a meal containing 40 g of protein from chicken
  Arms: Chicken

SUMMARY:
The aim of this study is to investigate the postprandial metabolic responses to plant-based meat alternatives made from different protein ingredients (pea, wheat or soy protein) in comparison to chicken in healthy adults. Therefore, young healthy subjects consume 4 test meals with 40 g of protein from pea protein, wheat protein, soy protein or chicken in a randomized order. In a postprandial period of 6 hours, parameters of protein, glucose and lipid metabolism (i.a. plasma amino acids), gastric emptying and hunger/satiety are analysed. It is assumed that the plasma amino acid profile after plant protein ingestion differs depending on protein source and in comparison to chicken protein.

DETAILED DESCRIPTION:
In a randomized crossover-design, 20 healthy women and men consume 4 test meals containing either 40 g of protein from plant-based meat alternatives (pea, wheat and soy protein extrudate) or chicken together with 1 g paracetamol, which is used as a marker for gastric emptying.

During a postprandial period of 6 hours parameters of protein metabolism (e.g. amino acids in plasma and urine), glucose metabolism (e.g. plasma glucose, serum insulin), lipid metabolism (serum triglycerides, total cholesterol , LDL cholesterol, HDL cholesterol, free fatty acids), serum uric acids, hunger- and satiety-associated gastrointestinal hormones (serum ghrelin, plasma GLP-1), and gastric emptying rate (based on plasma paracetamol) are analysed. Furthermore, subjective hunger/satiety and acceptance of the meals are assed using visual analogue scales. Each intervention arm will be separated by a washout period of at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* metabolically healthy
* normal weight (BMI: 18,5 - 24,9 kg/m2)
* written informed consent

Exclusion Criteria

* pregnancy, lactation
* hypo- or hypertension
* underweight or overweight/obesity
* food intolerances and allergies (especially soy, pea, wheat/gluten)
* malabsorption syndromes
* gastrointestinal diseases
* thyroid diseases
* diabetes mellitus type 1 and type 2
* impaired kidney or liver function
* anaemia
* blood coagulation disorders
* irregular menstrual cycle
* endometriosis, severe menstrual problems
* hormonal contraception
* regular use of medications (especially habitual use of paracetamol or medications that may interact with paracetamol)
* hypersensitivity to paracetamol
* body weight below 50 kg
* alcohol abuse
* glucose-6-phosphate dehydrogenase deficiency
* Gilbert's syndrome
* eating disorders (especially anorexia nervosa, bulimia nervosa)
* smoking
* participation in another study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Amino acid profile in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of amino acid profile in plasma (nmol/ml)

SECONDARY OUTCOMES:
Amino acid profile in urine | Postprandial period of 6 hours
  Analysis of amino acids in urine (nmol/mL)
Urea in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of urea (mg/dL) in blood
Nitrogen in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of nitrogen (mg/dL) in blood
Glucose in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of glucose (mmol/L) in blood
Insulin in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of insulin (pmol/L) in blood
C-peptide in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120 and 360 minutes)
  Analysis C-peptide (pg/ml) in blood
Glucagon in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of glucagon (pg/ml) in blood
Uric acid in blood | Postprandial period of 6 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of uric acid (mg/dL) in blood
Calcium in blood | Postprandial period of 6 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of calcium (mmol/l) in blood
Iron in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of iron (µg/l) in blood
Zinc in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of zinc (µg/l) in blood
Selenium in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of selenium (µg/l) in blood
Copper in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of copper (µg/l) in blood
Triglycerides in blood | Postprandial period of 6 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of triglycerides (mmol/l) in blood
Total cholesterol in blood | Postprandial period of 6 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of total cholesterol (mmol/l) in blood
LDL cholesterol in blood | Postprandial period of 6 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of LDL cholesterol (mmol/l) in blood
HDL cholesterol in blood | Postprandial period of 6 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of HDL cholesterol (mmol/l) in blood
Free fatty acids in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of free fatty acids (mmol/L) in blood
Gastric emptying rate | Postprandial period of 6 hours (Time points: fasting (0) and 30, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of gastric emptying rate based on paracetamol kinetics in blood (µg/mL)
Ghrelin in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240 and 360 minutes)
  Analysis of ghrelin (pg/mL) in blood
GLP-1 in blood | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180 and 360 minutes)
  Analysis of GLP-1 (pg/ml) in blood
Hunger/satiety and acceptance of the meals | Postprandial period of 6 hours (Time points: fasting (0) and 15, 30, 45, 60, 90, 120, 180, 240, 300 and 360 minutes)
  Assessment of subjective hunger/satiety and acceptance of the meals by validated visual analogue scale questionnaires (paper-pencil)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Egert, Prof PhD, Principal Investigator — University of Bonn, Institute of Nutritional and Food Sciences, Nutritional Physiology
Locations (1):
- University of Bonn, Institute of Nutritional and Food Sciences, Nutritional Physiology, Bonn, North Rhine-Westphalia, Germany